CLINICAL TRIAL: NCT01791894
Title: An Open-label, Biomarker Study of Arsenic Trioxide for the Treatment of Patients With Basal Cell Carcinoma
Brief Title: Arsenic Trioxide in Treating Patients With Basal Cell Carcinoma
Acronym: ATO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The V Foundation for Cancer Research (Other)
Responsible Party: Principal Investigator, Jean Yuh Tang, Associate Professor of Dermatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-26400; SKIN0015 (Other: OnCore)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Basal Cell Carcinoma of the Skin; Recurrent Skin Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (arsenic trioxide) (Experimental): Patients receive arsenic trioxide IV over 2 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox

SUMMARY:
This pilot clinical trial studies arsenic trioxide in treating patients with basal cell carcinoma. Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stop them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether administration of arsenic trioxide (ATO) to patients with basal cell carcinoma is associated with a reduction in Gli messenger ribonucleic acid (mRNA) and protein levels in tumor biopsy samples, when compared to baseline levels.

SECONDARY OBJECTIVES:

I. To determine whether there is evidence of tumor size reduction of ATO against basal cell carcinoma in humans.

OUTLINE:

Patients receive arsenic trioxide intravenously (IV) over 2 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
INCLUSION CRITERIA

* Basal cell carcinoma (BCC)
* Ineligible for curative locoregional treatment and have either progressed on, did not tolerate, unwilling to try or ineligible for investigational smoothened antagonist such as vismodegib (GDC 0449), XL 139 (BMS 833923), IPI- 926, LDE225 and PF-04449913
* Life expectancy estimate > 3 months
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits
* Corrected QT interval (QTC) by 12 lead electrocardiogram (EKG) < 450 msecs
* Serum potassium within normal limits
* Magnesium within normal limits
* Calcium within normal limits
* Ability to understand and the willingness to sign a written informed consent document
* Evaluable tumor and be potentially eligible for pre and post ATO tumor biopsy
* Receiving potassium wasting diuretics or amphotericin, while not excluded, must be noted to have theoretically increased arrhythmia risks with ATO

EXCLUSION CRITERIA

* Concurrent use of other Investigational agents
* Cardiac arrhythmias
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recurrent seizure history or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Results will be submitted to scientific journal for publication and shared at scientific meetings

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We will recruit from medical clinic and other physicians who treat metastatic BCC
Groups:
- IV ATO: 5 subjects will be treated with arsenic trioxide at 0.3 mg/kg daily via a 2 hour intravenous infusion for 5 days every 28 days (+/- 5 days) for a total of 3 cycles.
Period: Overall Study
Arm/Group | IV ATO
Started | 5
Completed | 4
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 5 patients with BCC who are not eligible for curative loco-regional treatment and have either progressed on, did not tolerate, unwilling to try or ineligible for investigational smoothened antagonist such as GDC 0449, XL 139 (BMS 833923), IPI- 926, LDE225 and PF-04449913 and fit the inclusion/exclusion criteria
Groups:
- Treatment (Arsenic Trioxide): arsenic trioxide IV over 2 hours on days 1-5. Courses repeat every 28 days
Arm/Group | Treatment (Arsenic Trioxide)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Biomarker (GLI2 Protein) Levels
Time Frame: baseline to day 33
Population: We recruited patients with biopsy-confirmed metastatic basal cell carcinoma who were had progressed on SMO inhibitors such as vismodegib (GDC 0449), IPI- 926, LEQ506 and LDE225.
Measure: Mean (Standard Deviation); unit: percentage decrease
Groups:
- Treatment (Arsenic Trioxide): Patients receive arsenic trioxide IV over 2 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  arsenic trioxide: Given IV
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Arsenic Trioxide)
Number analyzed (Participants) | 5
percentage decrease | 75 (11)

2. Secondary Outcome: Patients With Stable Disease Post Treatment
Description: Number of patients with stable disease post treatment by RECIST criteria
Time Frame: After 3 cycles of treatment (approx. 61 days)
Population: 4 patients completed 3 cycles of treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Arsenic Trioxide)
Number analyzed (Participants) | 4
participants | 3

3. Secondary Outcome: Patients With Progressive Disease Post Treatment by RECIST Criteria
Description: Patients with a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: After 3 treatment cycles (approx. 61 days)
Measure: Number; unit: participants
Arm/Group | IV ATO
Number analyzed (Participants) | 4
participants | 1

4. Secondary Outcome: Incidence of Grade 3/4 Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: Baseline to cycle 3
Measure: Number; unit: number of occurrences
Arm/Group | IV ATO
Number analyzed (Participants) | 5
number of occurrences | 2

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Treatment (Arsenic Trioxide)
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Arsenic Trioxide) (N=5)
grade 3 infection (Blood and lymphatic system disorders) | 1 (1) — Patient had a grade 3 infection after the cycle 3 arsenic trioxide infusion. Patient recovered after hospital admission and IV antibiotic treatment
grade 4 leukopenia (Blood and lymphatic system disorders) | 1 (1) — grade 4 leukopenia after the cycle 3 arsenic trioxide infusion. Patient recovered after hospital admission and IV antibiotic treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Arsenic Trioxide) (N=5)
grade 1 asymptomatic atrial flutter (Cardiac disorders) | 1 (1) — Patient 5discontinued treatment after the first cycle owing to grade 1 asymptomatic atrial flutter. He underwent repeated electrocardiography during a 1-week period, and the arrhythmia spontaneously resolved.
transaminitis (Investigations) | 1 (1) — grade 2 transaminitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No